CLINICAL TRIAL: NCT03038503
Title: What Should be the Next Vasopressor for Severe Septic Shock Patients? Methylene Blue or Terlipressin
Brief Title: What Should be the Next Vasopressor for Severe Septic Shock? Methylene Blue or Terlipressin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, munthana sundusadee, fellowship in department of pulmonary and critical care department, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ID 09-59-14
Record Dates: First submitted 2016-12-22; First posted 2017-01-31 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Septic Shock; Refractory Shock
Keywords: refractory septic shock; catecholamine resistance septic shock; terlipressin; methylene blue
MeSH Terms: conditions — Shock, Septic; Shock | interventions — Methylene Blue; Terlipressin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (No Intervention): standard care septic shock according sepsis bundles
- B (Experimental): after defined refractory shock (adequate fluid resuscitation + add NE>0.5 mcg/kg/min) add Methylene blue 1 mg/kg iv drip then 2 hr later drip 0.5 mg/kg/hr*4 hr (intervention add on to standard care)
  Interventions: Drug: Methylene Blue
- C (Experimental): after defined refractory shock (adequate fluid resuscitation + add NE>0.5 mcg/kg/min) add terlipressin 1 mg IV then repeated dose 20 min later if unstable BP (intervention add on to standard care)
  Interventions: Drug: Terlipressin

INTERVENTIONS:
Drug: Methylene Blue — after defined refractory shock (need NE>0.5 mcg/kg/min) add Methylene blue 1 mg/kg iv drip then 2 hr later drip 0.5 mg/kg/hr*4 hr (intervention add on to standard care)
  Arms: B
Drug: Terlipressin — after defined refractory shock (need NE>0.5 mcg/kg/min) add terlipressin 1 mg IV then repeated dose 20 min later if unstable BP (intervention add on to standard care)
  Arms: C

SUMMARY:
The ICU mortality rate of patients with septic shock was still high upto 54.1%.In first 6 hours of resuscitation, the goals of resuscitation in sepsis shock after adequate fluid resuscitation is MAP ≥65 mmHg. In refractory septic shock patient, prolong shock correlate with poor outcome due to multiple organ failure. Alternative vasopressor in septic shock with catecholamine resistance has been studied such as terlipressin, methylene blue

* Terlipressin (TP) mediate vasoconstriction via V1 receptors coupled to phospholipase C, and increases intracellular Ca2+ concentration
* Methylene blue (MB) directly inhibits nitric oxide synthase (NOS) by inhibit the enzyme guanylate cyclase (GC)

ELIGIBILITY:
Inclusion Criteria:

* Age >15 years old
* Diagnosis septic shock as SCCM/ACCP
* Refractory septic shock defined as hypotension although adequate fluid resuscitate and high dose vasopressor(NE >0.5 mcg/kg/min)
* Concent form

Exclusion Criteria:

* Known case G6PD deficiency
* Acute respiratory distress syndrome (ARDS)
* Hx of drug allergy MB, NE, terlipressin
* Hx of Raynaud's phenomenon, systemic sclerosis, PHT
* Known case coronary heart disease without treatment
* Current drug use serotonin reuptake inhibitors (SSRI), Serotonin and norepinephrine reuptake inhibitors (SNRIs)
* Reject to join project

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
mortality rate | 7 days
time to wean of vasopressor | through complete weaning off vasopressor, an average of 24 hours
ICU duration | through out off indication need ICU care, an average of 7 days

SECONDARY OUTCOMES:
hemodynamic parameter: Mean arterial pressure (mmHg) | every 30 min after start protocol up to 6 hr then every 1 hr up to 24 hours
  mmHg, A-line monitoring
hemodynamic parameter: lactate (mmol/l) | every 2 hr until 6 hr then every 4 hr until wean off vasopressor up to 24 hours
  mmol/l
hemodynamic parameter: urine output (ml) | every 2 hr until wean off vasopressor up to 24 hours
  ml

CONTACTS AND LOCATIONS:
Overall Officials: viratch tangsujaritvijit, MD, Study Chair — Mahidol University
Locations (1):
- Ramathibodi hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No